CLINICAL TRIAL: NCT07299916
Title: Transcranial Direct Current Stimulation (tDCS) and Immersive Virtual Reality Meditation(IVRM) for the Treatment of Anxiety Disorders: A Randomized Controlled Trial
Brief Title: Transcranial Direct Current Stimulation (tDCS) and Immersive Virtual Reality Meditation (IVRM) for the Treatment of Anxiety Disorders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lo Ka Ying, the hku mood team, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tDCS_anxiety
Record Dates: First submitted 2025-11-25; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; GAD
Keywords: immersive virtual reality meditation; Transcranial Direct Current Stimulation (tDCS); Augmentative treatment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At the start of each stimulation session, participants in both the active and sham tDCS groups underwent a current ramp-up from 0 to 2 mA; after this initial phase, the current was ramped back down to 0 mA exclusively for the sham group.
  Participants were informed that they might experience sensations such as tingling, headache, or mild burning during the first 30-60 seconds of stimulation. They were also told these sensations would likely subside over time as they acclimated to the procedure. This design ensured participants could not distinguish whether a reduction in side effects stemmed from habituation (active tDCS) or the current ramp-down (sham tDCS).
  Additionally, the tDCS device's stimulation mode was preconfigured by the principal investigator. This individual was not involved in delivering stimulation or measuring outcomes-two tasks handled by a research assistant who remained blinded to the stimulation mode.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS stimulation + IVRM (Experimental): Participants will receive 12 combined sessions (twice daily over 2 weeks), with each session being 20 minutes of active tDCS (delivering 2mA current, electrodes placed at left DLPFC (F3, anode) and right DLPFC (F4, cathode)) synchronized with immersive VR; a 20-minute interval between daily sessions
  Interventions: Device: tDCS +IVRM (Active stimulation)
- Sham tDCS stimulation + IVRM (Sham Comparator): Participants will receive 12 combined sessions (twice daily over 2 weeks), with each session being 20 minutes of sham tDCS synchronized with immersive VR; a 20-minute interval between daily sessions.
  In the sham condition, the current will be ramped up to 2mA within the first and last 30 seconds to mimic the sensation of stimulation, but then ramped down, with no current maintained at other times.
  Moreover, the stimulation mode of the tDCS device will be pre-set by a the principal investigator, who are not involved in the stimulation delivery or outcome measurements, both of which are conducted by a research assistant who are blinded to the stimulation mode.
  Interventions: Device: tDCS+IVRM (sham stimulation)

INTERVENTIONS:
Device: tDCS +IVRM (Active stimulation) — Participants will receive 12 combined sessions (twice daily over 2 weeks), with each session being 20 minutes of active tDCS (delivering 2mA current, electrodes placed at left DLPFC (F3, anode) and right DLPFC (F4, cathode)) synchronized with immersive VR; a 20-minute interval between daily sessions .The IVRM will employ guided meditation VR (Brainrise , France) ,as a technology based mindfulness based treatment, with standardised meditation scripts, using Oculus Rift VR headset. The current will be applied with the anode positioned left DLPFC, corresponding to area F3 in the international 10-20 system. The cathode will be applied at the right dPLFC, F4
  Arms: active tDCS stimulation + IVRM
Device: tDCS+IVRM (sham stimulation) — Participants will receive 12 sessions of sham tDCS stimulation paired with concurrent IVRM. Stimulation is delivered using a tDCS device (Soterix Medical), anodal stimulation at lDLPFC and cathodal stimulation at RFLPFC. The IVRM will employ guided meditation VR (Brainrise , France) ,as a technology based mindfulness based treatment, with standardised meditation scripts, using Oculus Rift VR headset. In the sham condition, the current will be ramped up to 2mA within the first and last 30 seconds to mimic the sensation of stimulation, but then ramped down, with no current maintained at other times.
  Arms: Sham tDCS stimulation + IVRM

SUMMARY:
The goal of this RCT is to evaluate the post-intervention (week 2) and 1-month post-intervention (week 6) of a 2-week intervention (12 sessions) of combined tDCS (a non-invasive brain stimulation method, with anodal stimulation over lDLPFC and cathodal stimulation over rDLPFC) and immersive virtual reality meditation (IVRM) on anxiety severity among individuals with anxiety disorders, as compared to sham group. We also assess the effects of the intervention on other secondary outcomes as compared to sham group, as well as the tolerability (how well people can handle it) and feasibility (how easy it is to carry out) of this combined intervention.

Exploratory analyses will examine physiological markers, such as heart rate variability (HRV), in relation to treatment response.

Participants will receive total 12 sessions of either active or sham tDCS on DLPFC paired with IVRM. The assessment will be blinded to assessors. No one (participants, researchers, assessors) will be revealed the group allocation. Sham tdcs applies the standard blinding protocol with 30 seconds of ramping up and ramping down periods.

Participants will:

Receive 12 total treatment sessions (twice a day for 2 weeks); each session is 20 minutes of tDCS (active or sham) plus IVRM. The IVRM uses HypnoVR® with 3D scenes (e.g., beach, forest) and 20-minute guided scripts meditation.Take a 20-minute break between the two daily sessions.

Complete assessments at three time points: baseline (before treatment, T0), right after the 2-week treatment (T1), and 1 month after treatment (T2). Assessments include anxiety tests (e.g., HAM-A, Beck Anxiety Inventory), adverse effect questionnaires (for tDCS and IVRM), and physiological checks (e.g., heart rate variability).

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-70 years;
* Diagnosed with Generalized Anxiety Disorder (GAD) or Mixed Anxiety and Depressive Disorder (MADD) or Major Depressive Disorder with prominent anxiety symptoms, according to the Structured Clinical Interview for DSM-5, Clinical Version (SCID-DSM-5, CV)
* Scored ≥ 8 (i.e., at least mild to moderate anxiety on the 14-item Hamilton Anxiety Rating Scale (HAM-A)) at screening;
* Right handedness;
* Stable dosage of antidepressants or other treatments for depression in recent 4 weeks; and
* Can read and write Chinese

Exclusion Criteria:

* History of significant head trauma, neurological disorders (e.g., epilepsy), seizures, or focal brain lesions;
* First degree relative with epilepsy, significant neurological illness or head trauma, endocrine disease;
* Concomitant unstable medical condition or major neurological conditions;
* Comorbid disorders listed in the DSM-V, e.g., schizophrenia, mental retardation, etc.;
* Current or history of alcohol or drug abuse;
* Inability to provide informed consent

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A)-14 items | Assessments are conducted at three time points: Baseline (Day 0, before the start of the intervention), post-intervention (Day 14, immediately after the 2-week combined tDCS-VR intervention), and 1-month post-intervention (Month 1, follow-up)
  The Hamilton Anxiety Rating Scale (HAM-A) is a 14-item clinician-rated tool used to assess the severity of anxiety symptoms, with scores ranging from 0 (minimum) to 56 (maximum); higher scores indicate more severe anxiety.

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Assessed at Baseline (Day 0), post-intervention (Day 1), and 1-month post-intervention (Month 1)
  The Beck Anxiety Inventory (BAI) is a 21-item self-report questionnaire designed to measure the severity of anxiety symptoms, with scores ranging from 0 to 63; higher scores indicate greater anxiety.
State-Trait Anxiety Inventory (STAI) | Assessed at Day 0, Day 14, and Month 1
  The State-Trait Anxiety Inventory (STAI) is a 40-item self-report measure that assesses two types of anxiety: state anxiety (temporary condition) and trait anxiety (general tendency), with scores ranging from 20 to 80 for each subscale; higher scores indicate greater anxiety.
Beck Depression Inventory (BDI) | Assessed at Day 0, Day 14, and Month 1
  The Beck Depression Inventory (BDI) is a 21-item self-report questionnaire used to assess the severity of depressive symptoms, with scores ranging from 0 to 63; higher scores indicate more severe depression.
Hamilton Depression Rating Scale (HDRS) | Assessed at Day 0, Day 14, and Month 1
  The Hamilton Depression Rating Scale (HDRS), also known as HAM-D, is a clinician-administered instrument commonly consisting of 17 items used to assess the severity of depressive symptoms, with scores typically ranging from 0 to 52; higher scores reflect more severe depression.
Montgomery-Åsberg Depression Rating Scale (MADRS) | Assessed in Day 0, Day 14, Month 1.
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-rated instrument consisting of 10 items designed to measure the severity of depressive symptoms, with scores ranging from 0 to 60; higher scores indicate more severe depression
The Hospital Anxiety and Depression Scale (HADS) | Assessed at Day 0
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report questionnaire designed to assess symptoms of anxiety (7 items) and depression (7 items) in non-psychiatric hospital settings, with each subscale scoring from 0 to 21; higher scores indicate greater symptom severity.
Somatic Symptom Scale (SSS-8) | Assessed Day 0, Day 14, Month 1
  The Somatic Symptom Scale - 8 (SSS-8) is an 8-item self-report questionnaire designed to assess the burden of somatic symptoms, with scores ranging from 0 to 32; higher scores indicate greater somatic symptom severity
Depression Anxiety Stress Scales (DASS-21) | Assessed at Day 0, Day 14, Month 1.
  The Depression Anxiety Stress Scales - 21 (DASS-21) is a 21-item self-report questionnaire designed to measure the severity of three related emotional states: depression, anxiety, and stress, with each subscale containing 7 items and scoring from 0 to 21; higher scores indicate greater symptom severity.
Perceived Stress Scale (PSS) | Assessed at Day 0, Day 14, Month 1.
  The Perceived Stress Scale (PSS) is a widely used self-report instrument consisting of 10 items that measure the degree to which individuals perceive situations in their life as stressful, with scores ranging from 0 to 40; higher scores indicate greater perceived stress.
Penn State Worry Questionnaire (PSWQ) | Assessed at Day 0, Day 14, Month 1.
  The Penn State Worry Questionnaire (PSWQ) is a 16-item self-report measure designed to assess the trait of worry, particularly its intensity and uncontrollability, with scores ranging from 16 to 80; higher scores indicate greater levels of pathological worry.
Multidimensional Fatigue Inventory (MFI) | Assessed at Day 0, Day 14, Month 1.
  The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report questionnaire designed to assess five dimensions of fatigue: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity, with each subscale scored from 4 to 20; higher scores indicate greater fatigue.
Short Form Health Survey (SF-6D) | Assessed at Day 0, Day 14, Month 1
  Short-form measure of health status from 6 dimensions.The SF-6D has been valued to generate utilities that reflect members of the public's preferences for health on the 0 to 1 utility scale (dead to full health) where values below zero indicate a health state that is considered worse than being dead. The lower the score, the more severe the disease.
Heart rate variability (HRV) | pre- and post-intervention time points; also during the intervention sessions
  By HeartMath Device and PULSAR android app
Visual Analog Scale (VAS) | Assessed at Day 14
  Two VASs items were used to measure motivation and willingness during intervention using a continuous scale. Each VAS contains a scale of 1 (minimum) to 10 (maximum). The total scores ranging from 2 to 20, with higher scores indicating more interest into the program and intervention
Adverse Effects Questionnaire for tDCS | Day 14 (post-assessment)
  Measure the adverse effects during the tDCS treatment period. 10 items of the potential adverse effects of tDCS. This instrument assesses the presence, severity , and perceived relatedness of ten common tDCS-associated sensations (e.g. itching, tingling headache, etc). Severity: For each present item, severity is graded on a 4-point scale (from 1-4): (No, Mild, Moderate, serious). The score ranges from 10-40. The higher the recorded score means the participants perceive more adverse effects from tDCS.
Simulator Sickness Questionnaire (SSQ) | At the end the intervention, Day 14 (Post-assessment)
  Record the Simulator Sickness for VR. There are 16 items, with each from 0-3 severity; The total score ranges from 0-48. Scores reflect the severity, with higher numbers meaning more sickness perceived by the participants.
Intervention tolerability and drop out rate | Post-assessment, Day 14.
  Measure the tolerability and drop out rate during the whole intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes